CLINICAL TRIAL: NCT04162132
Title: A Prospective Cohort Study of Contingency Management Using A Smartphone Application in Patients With Substance Use Disorder
Brief Title: Contingency Management Using Smartphone App in Patients With SUD
Status: Completed | Type: Observational
Sponsor: BrightView LLC (Industry)
Collaborators: DynamiCare Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 7135-SRyan
Record Dates: First submitted 2019-09-25; First posted 2019-11-14 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Substance Use Disorders
Keywords: contingency management; smartphone app; substance use disorder; outpatient addiction treatment; BrightView; DynamiCare
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DynamiCare group: Patients at Morgan Street location of BrightView who were given the DynamiCare smartphone app.
  Interventions: Device: Smartphone app
- Non-DynamiCare group: Patients at Colerain location of BrightView who were not given the DynamiCare smartphone app.

INTERVENTIONS:
Device: Smartphone app — Study procedures related to the DynamiCare Rewards intervention were conducted via smartphone. Research visits included collection of urine samples and medical exams. Participants assigned to the DynamiCare Rewards group received: 1) the app on their smartphone, 2) drug testing devices when indicated (pocket-sized breathalyzer), and a reloadable debit card for receiving the financial incentives (the PEX debit card). Global Positioning System (GPS) tracking was used to track whether patients had attended their scheduled appointments but was not used at any other times. All information was uploaded from the app onto the DynamiCare Analytics website, which treatment providers could view. The information reported was: attendance status of appointments, the status of all alcohol and drug testing, and incentives earned. Each patient's intervention period (period of time when they used the app) lasted four months from the date of their enrollment.
  Groups: DynamiCare group

SUMMARY:
The purpose of this research study is to test the acceptance and efficacy of a smartphone app (DynamiCare Rewards) for patients with substance use disorder (SUD) who are in active treatment and recovery at BrightView.

DETAILED DESCRIPTION:
The purpose of this research study was to test the acceptance and efficacy of a smartphone app (DynamiCare Rewards) for patients with substance use disorder (SUD) who are in active treatment and recovery at BrightView (www.brightviewhealth.com). Patients performed self-tracking of their recovery behavior (e.g., counseling attendance, abstinence from drugs and alcohol) addiction recovery behavior using the DynamiCare app, which follows Contingency Management (CM) model of incentivizing positive behavior.

CM is shown as a highly effective, evidence-based methodology for improving substance use disorder (SUD) outcomes. It does so by activating the brain's reward and inhibitory systems through both positive and negative reinforcement using immediate, concrete incentives in a progressive reinforcement schedule. CM involves setting frequent (>1/week), objective goals (usually abstinence or participation in treatment), which patients can achieve to earn tangible rewards (such as cash or vouchers). The DynamiCare smart phone app (iOS/Android) uses CM to incentivize patients to attend scheduled appointments and to submit negative alcohol and drug tests as they are rewarded for these behaviors. The intentions of this project were to assess whether use of the smartphone app as an add-on to treatment as usual could increase treatment retention, increase the percentage of appointments that were kept, and if substance use could be reduced for patients using the app.

Patients were enrolled in the study on a rolling basis from Jan 25, 2019 to March 29, 2019 until the desired cohort group # was reached (n=108). The intervention period (period of time when patients actually used the DynamiCare app) lasted four months from the date of their enrollment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Substance use disorder (SUD) as a primary diagnosis
* Have and use an Android or iOS smartphone with acceptable capability
* Are willing to participate in home testing and use of the smartphone
* Speak and read the English language adequately to understand smartphone commands and responses
* Are willing to be randomly assigned to receive treatment with or without the smartphone app as an added feature.

Exclusion Criteria:

• N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study focused on a population of 108 adult patients with a primary diagnosis of substance use disorder who were enrolled at a BrightView outpatient treatment center.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Attendance | 4 months
  The DynamiCare smart phone app was used to see whether the percentage of scheduled appointments could be increased by using the app. As measured by % of attendance of medical and clinical appointments compared to controls.
Substance Use | 4 months
  The DynamiCare smart phone app was used to see if use of the app could reduce substance use as measured by urine toxicology results. Measured percentage of patients using the app testing consistent only for prescribed substances in random clinical urine tests compared to controls.
Retention | 4 months
  The DynamiCare smart phone app was used to see if treatment retention could be increased when the app was added to treatment as usual. Measured as the percent of patients who are still active in the DynamiCare app and attending treatment sessions after 1, 2, 3, and 4 months compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Ryan, MD, MBA, Principal Investigator — President & CMO; Samin Rezania, PhD, Study Director — Director of Clinical Research
Locations (1):
- BrightView, Cincinnati, Ohio, United States

REFERENCES:
- See also: BrightView -- Outpatient addiction treatment center conducting the study — http://www.brightviewhealth.com
- See also: DynamiCare Health -- Maker of the smartphone app used in the study — http://dynamicarehealth.com

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04162132/Prot_000.pdf
  • Informed Consent Form (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04162132/ICF_001.pdf